CLINICAL TRIAL: NCT04602013
Title: A Prospective, Multi-center, Single-arm Clinical Study of Sintilimab Injection Combined With Concurrent Radiotherapy and Chemotherapy in the Treatment of Locally Advanced Esophageal Squamous Cell Carcinoma (IMCORT)
Brief Title: Sintilimab Injection Combined With Concurrent CCRT in Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: General Hospital of Ningxia Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Affiliated Hospital of Southwest Medical University (Other); Chongqing Three Gorges Central Hospital (Other)
Responsible Party: Principal Investigator, LI TAO, Section Head, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCHEC202007
Record Dates: First submitted 2020-08-24; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Locally Advanced Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma; chemoradiotherapy; immunity therapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sintilimab; Drug Therapy; Albumin-Bound Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy combined with chemoradiotherapy (Experimental): Immunotherapy combined with chemoradiotherapy
  1. Sintilimab Body weight <60kg: 3mg/kg IV Q3W; Body weight ≥60kg: 200mg IV Q3W.
  2. Chemotherapy drugs include cisplatin and albumin-bound paclitaxel for injection Paclitaxel for injection (albumin-bound type) dose: 3 dose groups (di=260 mg/m2, di-1=220 mg/m2, di-2=180 mg/m2).
     Dosing on the first day, one cycle every three weeks, a total of 2 cycles. Cisplatin (25mg/m2 IV D1-3 Q3W)
  3. Radiotherapy The total dose is 60-66 Gy, divided into 30-33 times (2.0 Gy/f, 5 f per week).
  Interventions: Drug: Sintilimab; Drug: Chemotherapy; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Sintilimab — Body weight <60kg: 3mg/kg IV Q3W; Body weight ≥60kg: 200mg IV Q3W. Every three weeks is a cycle
  Other Names: Sintilizumab
Drug: Chemotherapy — Chemotherapy drugs include cisplatin and albumin-bound paclitaxel for injection Paclitaxel for injection (albumin-bound type) dose: 3 dose groups (di=260 mg/m2, di-1=220 mg/m2, di-2=180 mg/m2).
  Dosing on the first day, one cycle every three weeks, a total of 2 cycles. Cisplatin (25mg/m2 IV D1-3 Q3W)
  Other Names: albumin-bound paclitaxel
Radiation: Radiation Therapy — The total dose is 60-66 Gy, divided into 30-33 times (2.0 Gy/f, 5 f per week).

SUMMARY:
This study evaluated the effectiveness and safety of sintilimab combined with cCRT in patients with locally advanced ESCC.

DETAILED DESCRIPTION:
This study evaluated the effectiveness and safety of sintilimab combined with cCRT in patients with locally advanced ESCC. The primary endpoint is PFS. Secondary points contains：ORR、OS、Qol.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or the legal representative of the patient can sign a written informed consent, and can understand and agree to follow the research requirements;
2. The age is between 18 and 75 when signing the informed consent;
3. Histologically diagnosed as locally advanced ESCC and suitable for CCRT, including: stage II-IVa (AJCC 8th edition [Rice et al., 2017]) inoperable ESCC patients (medical unsuitable for surgery or rejection of surgical intervention) Meet the criteria.
4. There are measurable and/or unmeasurable lesions that meet the definition of RECISTv1.1;
5. ECOG physical status ≤1;
6. Good organ function means that the laboratory test indicators obtained within 14 days before enrollment are as follows: a. Patients can achieve the following indicators without blood transfusion or growth factor treatment within 14 days before sample collection during the screening period i. Absolute neutrophils Cell count (ANC) ≥1.5×109/L ii. Platelet ≥100×109/L iii. Hemoglobin ≥90g/L b. Serum creatinine ≤1.5×ULN (upper limit of normal range), or through the epidemiological collaboration of chronic kidney disease Set of equation c. (Appendix 9) Estimated glomerular filtration rate ≥60mL/min/1.73m2 d. Serum total bilirubin≤1.5×ULN (The total bilirubin of patients with Gilbert syndrome must be ≤3× ULN). e. Aspartate aminotransferase and ALT<3×ULN.
7. The indicators for inactive/asymptomatic carriers, chronic or active HBV patients must meet: HBV deoxyribonucleic acid (DNA) during the screening period <500IU/mL (or 2500 copies/mL). Note: Patients with hepatitis B surface antigen positive or HBVDNA positive should be managed according to treatment guidelines. Patients receiving antiviral treatment during the screening period should have received treatment for >2 weeks before enrollment.
8. Women with fertility must voluntarily take effective contraceptive measures during the study period and within ≥120 days after the last administration of Sintilizumab, and the urine or serum pregnancy test results are negative within ≤7 days before enrollment 9. Not sterilized Of male subjects must voluntarily take effective contraceptive measures during the study period and ≥120 days after the last administration of Sintilimab.

Exclusion Criteria:

1. Have a history of fistula caused by primary tumor infiltration; 2. Patients with high risk of esophageal fistula or signs of esophageal perforation; 3. There is evidence of distant metastasis (M1 disease AJCC 8th edition [Rice et al., 2017]); 4. History of esophageal cancer surgery; 5. There are signs of severe malnutrition; 6. Pleural effusion, pericardial effusion or ascites that is clinically uncontrolled and requires repeated drainage or medical intervention (within 2 weeks before randomization); 7. Known to be intolerant or resistant to the chemotherapy specified in the trial protocol; 8. Have received radiotherapy, chemotherapy, targeted therapy, esophageal surgery or anti-PD-1, PD-L1, PD-L2 therapy or other tumor immunotherapy; 9. Patients with active autoimmune diseases or with a history of autoimmune diseases but may relapse Note: Patients with the following diseases are not excluded and can enter further screening: a. Controllable type I diabetes b. Hypothyroidism (only hormones are used) Alternative treatments can be controlled) c. Controllable celiac disease d. Skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, hair loss) e. Any other diseases that are not expected to recur if there is no external cause 10. Except for specific cancers under study in this study and locally recurring cancers that have been cured (eg, resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical or breast carcinoma in situ), before enrollment ≤2 years with other active malignant tumors 11. Any disease requiring systemic treatment with corticosteroids (dose>10mg/day of prednisone or equivalent doses of similar drugs) or other immunosuppressive agents within ≤14 days before randomization Note: Have used any of the following steroids currently or before Patients under the regimen are not excluded: a. Adrenaline replacement steroids (prednisone ≤10mg/day or equivalent dose of similar drugs) b. Local, ophthalmic, intra-articular, intranasal, or inhalation with minimal systemic absorption Corticosteroids c. Prophylactically short-term (≤7 days) use of corticosteroids (for example, to prevent allergy to contrast agents) or to treat non-autoimmune conditions (for example, delayed hypersensitivity reactions caused by contact with allergens) 12. ≤14 days before enrollment, uncontrolled diabetes, potassium, sodium, or corrected calcium laboratory test values >1 grade despite standard drug treatment, or hypoalbuminemia >3 grade 13.Have a history of interstitial lung disease, non-infectious pneumonia or uncontrolled systemic diseases, including pulmonary fibrosis, acute lung diseases, etc.

14. Severe chronic or active infection (including tuberculosis infection) that requires systemic antibacterial therapy, antifungal therapy or antiviral therapy in the 14 days before enrollment 15. Known history of HIV infection 16. Major surgery ≤28 days before enrollment Note: Minimally invasive surgery (such as central venous catheterization via peripheral venipuncture [PICC]) is not a major surgery.

17. Have received allogeneic stem cell transplantation or organ transplantation 18. There are any of the following cardiovascular risk factors: a. Cardiogenic chest pain ≤28 days before enrollment, defined as moderate pain that restricts daily appliance activities b. Symptomatic pulmonary embolism ≤28 days before enrollment c . Acute myocardial infarction occurred within ≤6 months before enrollment d. A history of heart failure reached New York Heart Association grade III or IV (Appendix 7) within ≤6 months before enrollment e. Before enrollment A ventricular arrhythmia event of grade ≥2 occurred within ≤6 months f. Cerebrovascular accident occurred within ≤6 months before enrollment g. ≤28 days before enrollment, despite the use of antihypertensive drugs, it has not been controlled Hypertension, namely systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg h. Syncope or seizure occurred ≤28 days before enrollment 19. History of severe hypersensitivity to other monoclonal antibodies or cisplatin or paclitaxel 20. Have received any chemotherapy, immunotherapy (such as interleukin, interferon, thymosin) or any research treatment within 14 days or 5 half-lives (whichever is shorter) before the first administration of the study drug 21. Have taken cancer control herbs within 14 days before the first dose of the study drug 22. Patients whose toxic and side effects caused by previous anti-tumor treatments have not returned to baseline or stable levels, unless they are considered to be AEs that are unlikely to bring safety risks (for example, hair loss, neuropathy, abnormal laboratory test values) 23. Live vaccines were vaccinated ≤28 days before enrollment. Note: Seasonal influenza vaccines are usually inactivated vaccines and are allowed to be used. Intranasal vaccines are live vaccines and are not allowed to be used.

24. There are underlying diseases (including abnormal laboratory test values) that are not conducive to the administration of study drugs, or have an impact on drug toxicity or the interpretation of AEs, or reduce or affect the subject's compliance to perform the study, alcohol or drug abuse, or rely.

25. At the same time participate in another therapeutic clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2020-10-11 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 3 years
  progression-free survival (PFS) refers to the time from enrollment to the first recording of disease progression as determined by RECISTv1.1, or to death due to any cause (whichever occurs first). PFS will be analyzed in the ITT analysis set.

SECONDARY OUTCOMES:
ORR | up to 3 years
  Objective response rate, according to RECISTv1.1, the proportion of patients with CR or PR was determined. If the patient has not undergone a post-baseline assessment, it is considered unremission.
Overall survival (OS | up to 5 years
  OS refers to the time from enrollment to the first recorded death due to any cause (whichever occurs first).
HRQoL | up to 3 years
  HRQoL uses EORTCQLQ-C30 to assess the overall health of patients. The post-baseline score of the treatment group was studied, and the score changes from the baseline were summarized descriptively.
HRQoL | up to 3 years
  HRQoL uses EORTCQLQ-OES18 to assess the overall health of patients. The post-baseline score of the treatment group was studied, and the score changes from the baseline were summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Li, Study Chair — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan Cancer Hospital & Institute, Chengdu, Sichuan, China